CLINICAL TRIAL: NCT02980198
Title: A Phase IIa, Single Blind, Randomized, Study to Evaluate the Safety, the Immunogenicity, and the Clinical and Biological Efficacy of IFNα-Kinoid (IFN-K) in Adult Subjects With Dermatomyositis
Brief Title: Study of IFN-K in Dermatomyositis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: reorganization proceedings with a potential risk of company liquidation
Sponsor: Neovacs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IFN-K-005-DM; 2016-000137-52 (EudraCT Number)
Record Dates: First submitted 2016-11-25; First posted 2016-12-02 (Estimated); Last update posted 2020-01-03 (Actual); Status verified 2019-12

CONDITIONS: Dermatomyositis
MeSH Terms: conditions — Dermatomyositis | interventions — montanide ISA 51

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IFN-Kinoid (Experimental): IFN-Kinoid + ISA 51
  Interventions: Biological: IFN-Kinoid; Other: ISA 51
- Placebo (Placebo Comparator): Placebo + ISA 51
  Interventions: Other: Placebo; Other: ISA 51

INTERVENTIONS:
Biological: IFN-Kinoid — IM administration
  Arms: IFN-Kinoid
Other: Placebo — IM administration
  Arms: Placebo
Other: ISA 51 — adjuvant

SUMMARY:
This study is a Proof of Concept study aiming to evaluate the production of anti-IFNα antibodies (immune response) in adult subjects with dermatomyositis

ELIGIBILITY:
Inclusion Criteria:

* Patient newly diagnosed or relapsing with "definite" or "probable" dermatomyositis based on ENMC criteria (2004)
* Patient requiring corticosteroids (CS) at a dose of 1 mg/Kg and ≤ 70 mg of prednisone equivalent/day or currently receiving CS at a dose of 1 mg/Kg and ≤ 70 mg of prednisone equivalent/day
* Is a male or female, aged between 18 and 65 years, inclusive, at the time of the screening visit
* study patient and his/her partner of child bearing potential has to use effective method of contraception

Exclusion Criteria:

* Is high-risk human papilloma virus (HPV) positive by (RT-PCR) on a cervical swab
* Has cytological abnormalities ≥ HSIL on a cervical swab
* Is positive for autoantibodies anti-NXP2, TIF1ɤ, MDA5 associated with severe pulmonary disease or anti-synthetase antibodies
* Is positive for any malignancy or has a history of any malignancy
* Has received IV pulse dose CS (≥ 250 mg prednisone equivalent/day)
* Has received intravenous immunoglobulin (IVIg)
* Has received potent immunosuppressive drugs such as cyclophosphamide, methotrexate, azathioprine, mycophenolate, cyclosporine A, oral tacrolimus
* Has received abatacept, anifrolumab, belimumab, TNF antagonists or another registered or investigational biological therapy
* Has received anti-B-cell therapy (e.g. rituximab, epratuzumab)
* Has received any live vaccine
* Has used any investigational or non-registered product , or any investigational or non-registered vaccine
* Has inflammatory joint or skin disease other than dermatomyositis that may interfere with study assessments
* Has frequent recurrences of oral or genital herpes simplex lesions
* Is at high risk of significant infection and/or has any current signs or symptoms of infection at entry or has received intravenous antibiotics

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-05-03 (Actual); Primary Completion 2019-12-11 (Actual); Study Completion 2019-12-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the expression of IFN-induced genes at Week 48 | Week 48

SECONDARY OUTCOMES:
Number of subjects with treatment related adverse events | Week 48
Total improvement score from IMAC Core Set Measures (CSM) following Aggarwal et al (2017) recommendations | Week 0, Week 12, Week 24, Week 36, Week 48
Others tools: Cutaneous Disease Area and Severity Index (CDASI) | Week 0, Week 12, Week 24, Week 36, Week 48
Others tools: Manual Muscle Testing (MMT5) | Week 0, Week 12, Week 24, Week 36, Week 48
Others tools: Accelerometer | Week 0, Week 12, Week 24, Week 36, Week 48
Others tools:Dermatology Life Quality Index (DLQI score) | Week 0, Week 12, Week 24, Week 36, Week 48
Immune response induced by IFN-K as measured by antibodies production | Week 48

CONTACTS AND LOCATIONS:
Locations (7):
- France (4):
  - Research site, Lille
  - Research site, Marseille
  - Research site, Paris
  - Research site, Strasbourg
- Charité - Universitätsmedizin Berlin Rudolf- Virchow- Haus, Berlin, Germany
- Research site, Padua, Italy
- Research site, Lausanne, Switzerland